CLINICAL TRIAL: NCT03568162
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of ISB 830 in Adult Subjects With Moderate to Severe Atopic Dermatitis.
Brief Title: Phase 2b Study to Evaluate the Efficacy and Safety of ISB 830 in Adults With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ichnos Sciences SA (Industry)
Collaborators: Glenmark Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBR 830-204; 2018-000783-29 (EudraCT Number)
Record Dates: First submitted 2018-05-31; First posted 2018-06-26 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-07

CONDITIONS: Moderate to Severe Atopic Dermatitis
Keywords: ISB 830, OX40, atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ISB 830 - Part 1 Group 1 (Experimental): Subcutaneous (SC) administration of ISB 830 as a loading dose, followed by SC maintenance dose of ISB 830.
  Interventions: Drug: ISB 830 - Part 1 Group 1
- ISB 830 - Part 1 Group 2 (Experimental): Subcutaneous (SC) administration of ISB 830 as a loading dose, followed by SC maintenance dose of ISB 830 or placebo.
  Interventions: Drug: ISB 830 - Part 1 Group 2
- ISB 830 - Part 1 Group 3 (Experimental): Subcutaneous (SC) administration of ISB 830 as a loading dose, followed by SC maintenance dose of ISB 830 or placebo.
  Interventions: Drug: ISB 830 - Part 1 Group 3
- Placebo - Part 1 Group 4 (Placebo Comparator): Subcutaneous (SC) administration of placebo, followed by SC maintenance dose of placebo.
  Interventions: Drug: Placebo - Part 1 Group 4
- ISB 830 - Part 2 Group 5 (Experimental): Subcutaneous (SC) administration of ISB 830 as a loading dose, followed by SC maintenance dose of ISB 830.
  Interventions: Drug: ISB 830 - Part 2 Group 5
- Placebo - Part 2 Group 6 (Placebo Comparator): Subcutaneous (SC) administration of placebo, followed by SC maintenance dose of placebo.
  Interventions: Drug: Placebo - Part 2 Group 6

INTERVENTIONS:
Drug: ISB 830 - Part 1 Group 1 — Subcutaneous injection (SC) every 2 weeks
  Arms: ISB 830 - Part 1 Group 1
Drug: ISB 830 - Part 1 Group 2 — Subcutaneous injection (SC) every 2 weeks
  Arms: ISB 830 - Part 1 Group 2
Drug: ISB 830 - Part 1 Group 3 — Subcutaneous injection (SC) every 2 weeks
  Arms: ISB 830 - Part 1 Group 3
Drug: Placebo - Part 1 Group 4 — Subcutaneous injection (SC) every 2 weeks
  Arms: Placebo - Part 1 Group 4
Drug: ISB 830 - Part 2 Group 5 — Subcutaneous injection (SC) every 2 weeks
  Arms: ISB 830 - Part 2 Group 5
Drug: Placebo - Part 2 Group 6 — Subcutaneous injection (SC) every 2 weeks
  Arms: Placebo - Part 2 Group 6

SUMMARY:
Phase 2b, randomized, double-blinded, placebo-controlled dose range finding study to evaluate the efficacy, safety and tolerability of ISB 830 in adults with moderate to severe atopic dermatitis. The study will be conducted in 2 Parts, with dosing Groups 1-4 comprising Part 1, and dosing Groups 5-6 comprising Part 2. All subjects will receive open-label ISB 830 after a 16 week blinded treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 years with physician diagnosis of atopic dermatitis for >1 year as defined by American Academy of Dermatology Consensus Criteria.
* Atopic dermatitis involvement of ≥10% of body surface area at screening and baseline.
* EASI score of ≥12 at screening or ≥16 at baseline.
* IGA score of ≥3 at screening and baseline (on the 0 to 4 IGA scale, in which 3 is moderate and 4 is severe)
* Baseline Pruritus Numerical Rating Scale (NRS) score for maximum itch intensity ≥3 over the previous 24 hours.

Exclusion Criteria:

* Pregnant or lactating women.
* Prior treatment with ISB 830
* Treatment with biologics
* Systemic corticosteroids, immunosuppressive/immunomodulatory drugs or phototherapy within 4 weeks of baseline
* Active chronic or acute infection requiring systemic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Acocella, MD, MBA, Study Director — Ichnos Sciences
Locations (83):
- United States (34):
  - Ichnos Investigational Site 129, Birmingham, Alabama
  - Ichnos Investigational Site 120, Clovis, California
  - Ichnos Investigational Site 105, Rolling Hills Estates, California
  - Ichnos Investigational Site 106, Bridgeport, Connecticut
  - Ichnos Investigational Site 146, Danbury, Connecticut
  - Ichnos Investigational Site 142, Brandon, Florida
  - Ichnos Investigational Site 143, Fort Myers, Florida
  - Ichnos Investigational Site 148, Lake City, Florida
  - Ichnos Investigational Site 141, Lake Worth, Florida
  - Ichnos Investigational Site 140, Miami, Florida
  - Ichnos Investigational Site 123, Miami, Florida
  - Ichnos Investigational Site 147, Ormond Beach, Florida
  - Ichnos Investigational site 101, Tampa, Florida
  - Ichnos Investigational Site 135, Tampa, Florida
  - Ichnos Investigational Site 115, Newnan, Georgia
  - Ichnos Investigational Site 139, Savannah, Georgia
  - Ichnos Investigational Site 112, Plainfield, Indiana
  - Ichnos Investigational Site 125, West Des Moines, Iowa
  - Ichnos Investigational Site109, New Orleans, Louisiana
  - Ichnos Investigational Site 126, St Louis, Missouri
  - Ichnos Investigational Site 144, Las Vegas, Nevada
  - Ichnos Investigational Site 117, Verona, New Jersey
  - Glenmark Investigational Site 102, Forest Hills, New York
  - Ichnos Investigational Site 114, Medford, Oregon
  - Ichnos Investigational Site 133, Hazleton, Pennsylvania
  - Ichnos Investigational Site 122, Philadelphia, Pennsylvania
  - Ichnos Investigational Site 132, Chattanooga, Tennessee
  - Ichnos Investigational Site 119, Houston, Texas
  - Ichnos Investigational Site 138, Pflugerville, Texas
  - Ichnos Investigational Site 116, San Antonio, Texas
  - Ichnos Investigational Site 110, Waco, Texas
  - Ichnos Investigational Site 103, Newport News, Virginia
  - Ichnos Investigational Site 131, Richmond, Virginia
  - Ichnos Investigational Site 136, Spokane, Washington
- Canada (9):
  - Ichnos Investigational Site 202, Calgary, Alberta
  - Ichnos Investigational Site 203, Surrey, British Columbia
  - Ichnos Investigational Site 207, Winnipeg, Manitoba
  - Ichnos Investigational Site 214, Hamilton, Ontario
  - Ichnos Investigational Site 204, Markham, Ontario
  - Ichnos Investigational Site 206, Ottawa, Ontario
  - Ichnos Investigational Site 208, Ottawa, Ontario
  - Ichnos Investigational Site 201, Richmond Hill, Ontario
  - Ichnos Investigational Site 211, Drummondville, Quebec
- Czechia (7):
  - Ichnos Investigational Site 404, Brno, Brno-město
  - Ichnos Investigational Site 402, Náchod, Královéhradecký kraj
  - Ichnos Investigational Site 403, Prague, Praha 3
  - Ichnos Investigational Site 401, Ostrava
  - Ichnos Investigational Site 405, Pardubice
  - Ichnos Investigational Site 407, Prague
  - Ichnos Investigational Site 406, Svitavy
- Germany (14):
  - Ichnos Investigational Site 313, Friedrichshafen, Baden-Wurttemberg
  - Ichnos Investigational Site 305, Langenau, Baden-Wurttemberg
  - Ichnos Investigational Site 311, Erlangen, Bavaria
  - Ichnos Investigational Site 314, Osnabrück, Lower Saxony
  - Ichnos Investigational Site 322, Bielefeld, North Rhine-Westphalia
  - Ichnos Investigational Site 318, Bochum, North Rhine-Westphalia
  - Ichnos Investigational Site 302, Dresden, Saxony
  - Ichnos Investigational Site 309, Dresden, Saxony
  - Ichnos Investigational Site 315, Lübeck, Schleswig-Holstein
  - Ichnos Investigational Site 319, Berlin
  - Ichnos Investigational Site 304, Berlin
  - Ichnos Investigational Site 326, Berlin
  - Ichnos Investigational Site 310, Hamburg
  - Ichnos Investigational Site 308, Hamburg
- Poland (19):
  - Ichnos Investigational Site 518, Poznan, Greater Poland Voivodeship
  - Ichnos Investigational Site 514, Poznan, Greater Poland Voivodeship
  - Ichnos Investigational Site 502, Krakow, Lesser Poland Voivodeship
  - Ichnos Investigational Site 511, Krakow, Lesser Poland Voivodeship
  - Ichnos Investigational Site 510, Krakow, Lesser Poland Voivodeship
  - Ichnos Investigational Site 501, Krakow, Lesser Poland Voivodeship
  - Ichnos Investigational Site 504, Wroclaw, Lower Silesian Voivodeship
  - Ichnos Investigational Site 509, Warsaw, Masovian Voivodeship
  - Ichnos Investigational Site 521, Warsaw, Masovian Voivodeship
  - Ichnos Investigational Site 512, Warsaw, Masovian Voivodeship
  - Ichnos Investigational Site 506, Warsaw, Masovian Voivodeship
  - Ichnos Investigational Site 517, Iwonicz-Zdrój, Podkarpackie Voivodeship
  - Ichnos Investigational Site 519, Gdynia, Pomeranian Voivodeship
  - Ichnos Investigational Site 520, Gdynia, Pomeranian Voivodeship
  - Ichnos Investigational Site 513, Szczecin, West Pomeranian Voivodeship
  - Ichnos Investigational Site 503, Katowice
  - Ichnos Investigational Site 505, Krakow
  - Ichnos Investigational Site 508, Skarżysko-Kamienna
  - Ichnos Investigational Site 507, Warsaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 4 phases: a Screening phase (28 days before randomization), a Blinded Treatment Phase (up to Week 16), an Open-label Treatment Phase (Week 16 to Week 54), and a Follow-up Phase (Week 54 to Week 66)
Pre-assignment Details: During Blinded Treatment Phase, participants received placebo-controlled treatment with ISB 830 administered subcutaneously (SC) for 16 weeks at different dose levels. During the Open-label Treatment Phase, participants received treatment with ISB 830 administered SC every other week (q2w) for 38 weeks.
Groups:
- ISB 830 300 mg q2w: Blinded Treatment Phase: ISB 830 administered at dose of 600 mg via SC injection (2 × 300 mg) on Day 1, followed by ISB 830 administered at dose of 300 mg (1 × 300 mg) via SC injection every 2 weeks (q2w) starting from Day 15 (Week 2) up to Week 14.
  Open-label Treatment Phase: ISB 830 administered at dose of 300 mg (1 × 300 mg) via SC injection q2w starting from Week 16 up to Week 52 (or until participant withdrawal). Participants were followed up for 12 weeks after treatment discontinuation, maximum up to Week 66.
- ISB 830 300 mg q4w: Blinded Treatment Phase: ISB 830 administered at dose of 600 mg via SC injection (2 × 300 mg) on Day 1, followed by ISB 830 administered at dose of 300 mg (1 × 300 mg) via SC injection every 4 weeks (q4w) starting from Day 29 (Week 4) up to Week 12 and placebo administered via SC injection q4w starting from Day 15 (Week 2) up to Week 14.
  Open-label Treatment Phase: ISB 830 administered at dose of 300 mg (1 × 300 mg) via SC injection q2w starting from Week 16 up to Week 52 (or until participant withdrawal). Participants were followed up for 12 weeks after treatment discontinuation, maximum up to Week 66.
- ISB 830 75 mg q4w: Blinded Treatment Phase: ISB 830 administered at dose of 150 mg via SC injection (2 × 75 mg) on Day 1, followed by ISB 830 administered at dose of 75 mg (1 × 75 mg) via SC injection q4w starting from Day 29 (Week 4) up to Week 12 and placebo administered via SC injection q4w starting from Day 15 (Week 2) up to Week 14.
  Open-label Treatment Phase: ISB 830 administered at dose of 300 mg (1 × 300 mg) via SC injection q2w starting from Week 16 up to Week 52 (or until participant withdrawal). Participants were followed up for 12 weeks after treatment discontinuation, maximum up to Week 66.
- Placebo - 1: Blinded Treatment Phase: Placebo administered via SC injection (2 injections) q2w starting from Day 1 up to Week 14.
  Open-label Treatment Phase: ISB 830 administered at dose of 300 mg (1 × 300 mg) via SC injection q2w starting from Week 16 up to Week 52 (or until participant withdrawal). Participants were followed up for 12 weeks after treatment discontinuation, maximum up to Week 66.
- ISB 830 600 mg q2w: Blinded Treatment Phase: ISB 830 administered at dose of 1200 mg via SC injection (4 × 300 mg) on Day 1, followed by ISB 830 administered at dose of 600 mg (2 × 300 mg) via SC injection q2w starting from Day 15 (Week 2) up to Week 14.
  Open-label Treatment Phase: ISB 830 administered at dose of 600 mg (2 × 300 mg) via SC injection q2w starting from Week 16 up to Week 52 (or until participant withdrawal). Participants were followed up for 12 weeks after treatment discontinuation, maximum up to Week 66.
- Placebo - 2: Blinded Treatment Phase: Placebo administered via SC injection (4 injections) q2w starting from Day 1 up to Week 14.
  Open-label Treatment Phase: ISB 830 administered at dose of 600 mg (2 × 300 mg) via SC injection q2w starting from Week 16 up to Week 52 (or until participant withdrawal). Participants were followed up for 12 weeks after treatment discontinuation, maximum up to Week 66.
Period: Overall Study
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Started | 76 | 80 | 77 | 80 | 75 | 74
Completed | 54 | 57 | 42 | 50 | 61 | 60
Not Completed | 22 | 23 | 35 | 30 | 14 | 14
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 2 | 4 | 2 | 3 | 2
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 15 | 15 | 26 | 22 | 6 | 9
Not completed — Others | 3 | 4 | 1 | 4 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of study medication. Participants were analyzed according to the treatment group assigned. Two participants randomized to ISB 830 300 mg q4w group discontinued study without receiving any study drug and were excluded from FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2 | Total
Number analyzed (Participants) | 76 | 78 | 77 | 80 | 75 | 74 | 460
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (13.10) | 36.6 (14.77) | 38.4 (16.87) | 36.3 (13.05) | 37.9 (13.31) | 36.0 (13.75) | 37.55 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 44 | 41 | 44 | 37 | 47 | 245
  Male | 44 | 34 | 36 | 36 | 38 | 27 | 215
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 2 | 2 | 3 | 0 | 15
  Not Hispanic or Latino | 71 | 75 | 75 | 78 | 72 | 73 | 444
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 4 | 4 | 7 | 2 | 1 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 14 | 6 | 15 | 6 | 4 | 58
  White | 58 | 59 | 65 | 58 | 66 | 69 | 375
  More than one race | 0 | 1 | 2 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.72 (7.538) | 27.49 (6.167) | 26.32 (6.199) | 27.20 (6.608) | 26.03 (5.167) | 26.50 (5.434) | 27.05 (6.27)
Baseline Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: units on a scale] — In EASI, four disease characteristics of atopic dermatitis (AD) (erythema, edema/papulation, excoriation, and lichenification) are assessed for severity. The EASI score ranges from 0 to 72 points, with the highest score indicating worse severity of AD.
  units on a scale | 30.42 (14.110) | 33.84 (14.910) | 28.42 (11.602) | 30.65 (13.173) | 29.86 (13.223) | 31.81 (14.340) | 30.84 (13.630)
Baseline Severity scoring of Atopic Dermatitis (SCORAD) Score [Mean (Standard Deviation); unit: units on a scale] — SCORAD is a composite severity index score. A SCORAD score ranges from 0 (no AD present) to 103 (severe).
  units on a scale | 67.50 (14.325) | 69.09 (14.284) | 66.22 (12.408) | 66.12 (12.658) | 66.40 (12.300) | 67.66 (13.560) | 67.16 (13.250)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Clinical Score at Week 16
Description: In EASI, four disease characteristics of atopic dermatitis (AD) (erythema, edema/papulation, excoriation, and lichenification) are assessed for severity on a scale of 0 (absent), 1 (mild), 2 (moderate), 3 (severe). The scores are added up for each of the four body regions (Head and neck, trunk, arms, and legs). The assigned percentages of body surface area (BSA) for each section of the body are 10% for head and neck, 20% for arms, 30% for trunk, and 40% for legs. Each subtotal score is multiplied by the BSA represented by that region. In addition, an area score of 0 to 6 is assigned for each body region, depending on the percentage of AD-affected skin in that area: 0 (none), 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). Each of the body area scores are multiplied by the area affected. The resulting EASI score ranges from 0 to 72 points, with the highest score indicating worse severity of AD.
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of study medication. Participants were analyzed according to the treatment group assigned. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 51 | 45 | 39 | 42 | 53 | 51
percentage change | -57.589 (36.2014) | -56.734 (32.5395) | -38.099 (39.6857) | -42.142 (38.1945) | -59.737 (27.1176) | -43.252 (41.2404)
Statistical Analysis 1: Comparison: ISB 830 300 mg q2w vs Placebo - 1; Test type: Superiority — The analysis was conducted using a mixed model for repeated measures (MMRM) model for percent change from baseline in EASI with the corresponding baseline value as covariate, and treatment group, region, disease severity, visit as fixed effect factors, and interactions of treatment-by-visit, baseline-by-visit; p = 0.008, Mixed Models Analysis; LS Mean Difference = -20.192, 95% CI 2-sided [-34.944 to 5.439], Standard Error of Mean 7.4781 — A linear contrast was used to estimate the treatment difference
Statistical Analysis 2: Comparison: ISB 830 300 mg q4w vs Placebo - 1; Test type: Superiority — The analysis was conducted using a MMRM model for percent change from baseline in EASI with the corresponding baseline value as covariate, and treatment group, region, disease severity, visit as fixed effect factors, and interactions of treatment-by-visit, baseline-by-visit; p = 0.061, Mixed Models Analysis; LS Mean Difference = -14.439, 95% CI 2-sided [-29.552 to 0.674], Standard Error of Mean 7.6622 — A linear contrast was used to estimate the treatment difference
Statistical Analysis 3: Comparison: ISB 830 75 mg q4w vs Placebo - 1; Test type: Superiority — The analysis was conducted using a mixed MMRM model for percent change from baseline in EASI with the corresponding baseline value as covariate, and treatment group, region, disease severity, visit as fixed effect factors, and interactions of treatment-by-visit, baseline-by-visit; p = 0.691, Mixed Models Analysis; LS Mean Difference = 3.144, 95% CI 2-sided [-12.410 to 18.698], Standard Error of Mean 7.8864 — A linear contrast was used to estimate the treatment difference
Statistical Analysis 4: Comparison: ISB 830 600 mg q2w vs Placebo - 2; The analysis was conducted using a MMRM model for percent change from baseline in EASI with the corresponding baseline value as covariate, and treatment group, region, disease severity, visit as fixed effect factors, and interactions of treatment-by-visit, baseline-by-visit; Test type: Superiority; p = 0.008, Mixed Models Analysis; LS Mean Difference = -17.199, 95% CI 2-sided [-29.895 to -4.503], Standard Error of Mean 6.4090 — A linear contrast was used to estimate the treatment difference

2. Secondary Outcome: Percentage of Participants Achieving a 75% Reduction From Baseline in EASI Score (EASI-75) at Week 16
Description: In EASI, 4 disease characteristics of AD are assessed for severity on a scale of 0 (absent), 1 (mild), 2 (moderate), 3 (severe). The scores are added up for each of the 4 body regions (Head and neck, trunk, arms, and legs). The assigned percentages of BSA for each section of the body are 10% for head and neck, 20% for arms, 30% for trunk, and 40% for legs. Each subtotal score is multiplied by the BSA represented by that region. In addition, an area score of 0 to 6 is assigned for each body region, depending on the percentage of AD-affected skin: 0 (none), 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). Each of the body area scores are multiplied by the area affected. The resulting EASI score ranges from 0 to 72 points, with the highest score indicating worse severity of AD.
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of study medication. Participants were analyzed according to the treatment group assigned. Any participant who received a rescue medication for AD during Part 1, had missed Week 16 assessment, or withdrew before Week 16 was considered Non-responder.
Measure: Number; unit: percentage of participants
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 76 | 78 | 77 | 80 | 75 | 74
percentage of participants | 23.7 | 20.5 | 11.7 | 11.3 | 25.3 | 18.9

3. Secondary Outcome: Percentage of Participants Achieving Both Investigator's Global Assessment (IGA) Clinical Score of 0 or 1 and an IGA Reduction From Baseline of ≥ 2 Points at Week 16
Description: The IGA is an assessment scale used in clinical studies to determine severity of AD based on a 5-point scale ranging from 0 (clear) to 4 (severe/very severe).
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 76 | 78 | 77 | 80 | 75 | 74
percentage of participants | 13.2 | 10.3 | 6.5 | 5.0 | 12.0 | 5.4

4. Secondary Outcome: Percentage of Participants With Improvement (Reduction) in Pruritus Numerical Rating Scale (NRS) Score of ≥ 4 From Baseline at Week 16
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Pruritus NRS was analyzed based on weekly rolling averages of daily scores.
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of study medication. Participants were analyzed according to the treatment group assigned. Any participant who received a rescue medication for AD during Part 1, had missed Week 16 assessment or withdrew before Week 16 was considered Non-responder.
Measure: Number; unit: percentage of participants
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 76 | 78 | 77 | 80 | 75 | 74
percentage of participants | 7.9 | 11.5 | 5.2 | 10.0 | 13.3 | 9.5

5. Secondary Outcome: Percentage of Participants Achieving a 50% Reduction From Baseline in EASI Score (EASI-50) at Week 16
Description: as for outcome 2
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of study medication. Participants were analyzed according to the treatment group assigned. Any participant who received a rescue medication for AD during Part 1, had missing Week 16 assessment, or withdrew before Week 16 was considered Nonresponder
Measure: Number; unit: percentage of participants
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 76 | 78 | 77 | 80 | 75 | 74
percentage of participants | 48.7 | 34.6 | 27.3 | 27.5 | 44.0 | 33.8

6. Secondary Outcome: Percent Change From Baseline in SCORAD Score at Week 16
Description: SCORAD (Severity scoring of Atopic Dermatitis) is composite severity index comprising a) the amount/extent of BSA affected; b) subjective symptom visual analog assessments for pruritis ( 0 [no itching] to 3 [severe itching]) and sleep disturbance (0 [no sleep disturbance] to 3 [severe sleep disturbance]); and c) 6 disease intensity assessments [dryness/scaling, erythema, induration/papulation, excoriation, lichenification and oozing/weeping/crusting, each graded from 0 to (none) to 3 (severe). A SCORAD score ranges from 0 (no AD present) to 103 (severe).
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 51 | 45 | 39 | 42 | 53 | 51
percentage change | -26.519 (18.1662) | -26.108 (21.4476) | -18.405 (15.8756) | -19.440 (17.4296) | -27.401 (14.4471) | -18.847 (14.4472)

7. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a 10-item validated questionnaire used to assess the impact of AD disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much). Item scores are added to provide a total score, ranging from 0 to 30, with higher scores indicating greater impairment of QoL.
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of study medication. Participants were analyzed according to the treatment group assigned. Here, 'Overall Number of Participants Analyzed' signifies the number of participants analyzed for this outcome measure and 'Number Analyzed' signifies the number of participants analyzed at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 76 | 78 | 77 | 80 | 75 | 74
units on a scale
  Baseline | 15.2 (6.80) | 15.4 (7.14) | 14.3 (7.18) | 14.3 (6.77) | 14.1 (6.02) | 14.7 (6.78)
  Change at Week 16: number analyzed (Participants) | 51 | 44 | 39 | 42 | 52 | 51
  Change at Week 16 | -7.3 (7.58) | -6.7 (6.16) | -4.1 (6.13) | -4.7 (7.00) | -6.6 (6.19) | -5.5 (5.10)

8. Secondary Outcome: Change From Baseline in Global Individual Signs Score (GISS) at Week 16
Description: GISS assesses AD lesions for erythema, excoriations, lichenification and infiltration/papulation. Each component is rated on a global basis (over the entire body surface rather than region) using a 4-point scale (0=none, 1=mild, 2=moderate, and 3=severe) according to the EASI grading severity. Total score ranges from 0 to 12 (no disease to most severe disease, respectively).
Time Frame: Baseline, Week 16
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 76 | 78 | 77 | 80 | 75 | 74
units on a scale
  Baseline | 9.1 (1.81) | 9.4 (1.71) | 9.1 (1.71) | 8.9 (1.77) | 9.0 (1.66) | 8.9 (1.63)
  Change at Week 16: number analyzed (Participants) | 51 | 45 | 39 | 42 | 53 | 51
  Change at Week 16 | -3.4 (2.52) | -3.2 (2.81) | -2.4 (2.52) | -2.2 (2.49) | -3.5 (2.52) | -2.3 (2.21)

9. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Subscale Scores at Week 16
Description: The HADS is a 14-item questionnaire, with 7 items related to anxiety (HADS-A) and 7 items related to depression (HADS-D). Each item is scored from 0 to 3; scores for each subscale range from 0 to 21, with higher scores indicating more distress. For each subscale, scores 7 or lower are considered normal, 8 to 10 are borderline, and 11 or higher indicate clinical anxiety or depression.
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of study medication. Participants were analyzed according to the treatment group assigned. Here, 'Overall Number of Participants Analyzed' signifies the number of participants analyzed for this outcome measure and 'Number Analyzed' signifies the number of participants analyzed for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 76 | 78 | 77 | 80 | 75 | 74
units on a scale
  HADS-A Baseline | 6.1 (4.47) | 6.1 (4.82) | 6.1 (4.15) | 6.2 (3.74) | 6.0 (4.41) | 6.7 (4.12)
  HADS-D Baseline | 4.3 (3.90) | 4.8 (4.38) | 4.9 (4.19) | 4.2 (3.16) | 4.7 (3.81) | 5.0 (4.26)
  HADS-A Change at Week 16: number analyzed (Participants) | 51 | 44 | 39 | 42 | 52 | 51
  HADS-A Change at Week 16 | -1.8 (3.34) | -0.9 (3.54) | -1.0 (3.16) | -0.8 (3.39) | -1.8 (3.80) | -1.9 (3.85)
  HADS-D Change at Week 16: number analyzed (Participants) | 51 | 44 | 39 | 42 | 52 | 51
  HADS-D Change at Week 16 | -1.1 (2.62) | -1.0 (4.05) | -0.6 (2.58) | -0.1 (2.62) | -0.9 (3.60) | -1.2 (2.97)

10. Secondary Outcome: Change From Baseline in Patient-Oriented Eczema Measure (POEM) at Week 16
Description: The POEM is a 7-item, validated questionnaire used to assess disease symptoms in both children and adults. Participants respond to 7 questions, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency of occurrence during the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores are added to provide a total score ranging from 0 (clear) to 28 (very severe atopic eczema).
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of study medication. Participants were analyzed according to the treatment group assigned. Here, 'Overall Number of Participants Analyzed' signifies the number of participants analyzed for this outcome measure and 'Number Analyzed' signifies the number of participants analyzed for specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 76 | 78 | 77 | 80 | 75 | 74
units on a scale
  Baseline | 20.2 (5.78) | 20.9 (5.56) | 19.8 (5.27) | 21.2 (5.40) | 20.7 (4.63) | 21.1 (4.79)
  Change at Week 16: number analyzed (Participants) | 51 | 44 | 39 | 42 | 52 | 51
  Change at Week 16 | -7.1 (6.44) | -4.8 (8.79) | -3.8 (6.51) | -5.0 (6.94) | -7.0 (7.37) | -5.5 (7.33)

11. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Disease and Treatment at Week 16
Description: For PGA of disease, participants rated their overall wellbeing on a 5-point Likert scale from 0 (poor) to 4 (excellent). Participants were asked: "Considering all the ways in which your disease affects you, indicate how well you are doing." Response choices were: "Poor"; "Fair"; "Good"; "Very Good"; "Excellent." For PGA of treatment, participants rated their satisfaction with the study treatment on a 5-point Likert scale from 0 (poor) to 4 (excellent). Subjects were asked: "How would you rate the way your disease responded to the study medication?" Response choices were: "Poor"; "Fair"; "Good"; "Very Good"; "Excellent".
Time Frame: Baseline, Week 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 76 | 78 | 77 | 80 | 75 | 74
units on a scale
  PGA of Disease Baseline | 2.0 (0.89) | 1.9 (0.84) | 2.1 (0.97) | 1.9 (0.79) | 2.0 (0.76) | 2.1 (0.92)
  PGA of Treatment Baseline: number analyzed (Participants) | 70 | 63 | 65 | 69 | 67 | 67
  PGA of Treatment Baseline | 2.1 (0.98) | 2.0 (1.07) | 2.1 (0.98) | 2.0 (1.05) | 2.2 (1.02) | 1.9 (1.03)
  PGA of Disease Change at Week 16: number analyzed (Participants) | 51 | 44 | 39 | 42 | 52 | 51
  PGA of Disease Change at Week 16 | 1.1 (0.98) | 1.2 (1.17) | 0.8 (0.80) | 1.1 (0.97) | 1.1 (0.88) | 0.8 (0.83)
  PGA of Treatment Change at Week 16: number analyzed (Participants) | 50 | 41 | 37 | 41 | 52 | 49
  PGA of Treatment Change at Week 16 | 0.9 (0.87) | 1.1 (0.98) | 0.7 (0.75) | 0.7 (0.84) | 1.0 (0.88) | 0.7 (0.92)

12. Secondary Outcome: Percentage Change From Baseline in PGA of Disease and Treatment at Week 16
Description: as for outcome 11
Time Frame: Baseline, Week 16
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of study medication. Participants were analyzed according to the treatment group assigned. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure and 'Number Analyzed' signifies the number of participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 51 | 44 | 39 | 42 | 52 | 51
percentage change
  PGA of Disease: Percent Change at Week 16 | 72.2 (93.51) | 73.3 (114.18) | 33.3 (87.25) | 76.2 (101.89) | 69.2 (92.85) | 40.4 (76.89)
  PGA of Treatment: Percent Change at Week 16: number analyzed (Participants) | 50 | 41 | 37 | 41 | 52 | 49
  PGA of Treatment: Percent Change at Week 16 | 42.3 (75.61) | 50.6 (97.24) | 16.0 (64.62) | 21.3 (56.76) | 55.0 (93.81) | 15.2 (61.29)

13. Secondary Outcome: Number of Missed Work or School Days at Week 16
Description: Participants who were employed or enrolled in school were asked to report the number of sick leave and/or missed school days due to AD (eg, versus due to an accident) in the last 4 weeks.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 44 | 35 | 31 | 32 | 34 | 38
days | 1.2 (3.73) | 0.5 (0.92) | 0.5 (1.26) | 0.5 (1.29) | 4.9 (14.92) | 1.4 (5.31)

14. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of ISB 830
Description: Cmax is the maximum concentration of ISB 830 observed in serum
Time Frame: Predose (within 15 minutes prior to dose), 4, 24, 96, 120, 168, and 336 hours postdose on Day 1 and predose (within 15 minutes prior to dose), 4, 24, 96, 120, and 168 hours postdose on Day 85
Population: Pharmacokinetic Analysis Set (PKAS) included all participants who received at least 1 dose of ISB 830, did not had any major protocol deviation affecting pharmacokinetic (PK), and for whom at least 1 sample with detectable plasma concentration with known time of dosing and the time of sampling was available. 'Overall Number of Participants Analyzed' = number of participants evaluable for this outcome measure; 'Number Analyzed' = number of participants evaluable at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliters (µg/mL)
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | ISB 830 600 mg q2w
Number analyzed (Participants) | 12 | 14 | 14 | 3
micrograms per milliliters (µg/mL)
  Day 1 | 46.98 (46.5) | 49.95 (33.1) | 16.62 (32.6) | 92.84 (12.3)
  Day 85: number analyzed (Participants) | 11 | 13 | 10 | 2
  Day 85 | 52.33 (45.8) | 31.20 (60.4) | 8.8 (73.6) | 144.80 (6.8)

15. Secondary Outcome: Area Under Curve From Time Zero to the End of Dosing Interval (AUC0-tau)
Description: AUC0-tau is the area under the curve from time zero to the end of the dosing interval of ISB 830.
Time Frame: Predose (within 15 minutes prior to dose), 4, 24, 96, 120, 168, and 336 hours postdose on Day 1 and predose (within 15 minutes prior to dose), and at 4, 24, 96, 120, 168 hours postdose on Day 85
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | ISB 830 600 mg q2w
Number analyzed (Participants) | 12 | 14 | 13 | 2
h*µg/mL
  Day 1: number analyzed (Participants) | 12 | 14 | 13 | 1
  Day 1 | 12170 (49.9) | 20340 (34.1) | 6671 (40.2) | 26930
  Day 85: number analyzed (Participants) | 10 | 13 | 7 | 2
  Day 85 | 12990 (40.3) | 13120 (49.5) | 3448 (97.8) | 39420 (2.6)

16. Secondary Outcome: Percentage of Participants With Anti-Drug Antibody (ADA) at Week 16
Description: Participants with ADA were those with at least 1 treatment-induced or treatment-boosted ADA-positive sample at any time during the treatment or follow-up observation period (up to Week 16). Treatment-emergent ADA referred to percentage of the total number of evaluable participants who were ADA-negative at baseline but developed ADA following biologic drug administration. Treatment-boosted ADA referred to percentage of the total number of evaluable participants who were ADA positive at baseline with at least 4-fold increase in ADA titer after biologic drug administration.
Time Frame: Baseline through Week 16
Population: Safety Analysis Set (SAS) included all participants who were randomized and received at least 1 dose of study medication. Participants were analyzed according to the treatment they received. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 | ISB 830 600 mg q2w | Placebo - 2
Number analyzed (Participants) | 75 | 77 | 77 | 79 | 75 | 74
percentage of participants | 13.3 | 29.9 | 50.6 | 5.1 | 10.7 | 6.8

ADVERSE EVENTS:
Time Frame: Up to Week 54
Description: An adverse event (AE) is defined as any untoward medical occurrence and does not necessarily have to have causal relationship with the study medication. An AE can therefore be an unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease, which is a change from baseline and is temporally associated with the use of the study medication, whether or not it is considered related to the study medication
Groups:
- Placebo - 1 (Blinded): Blinded Treatment Phase: Placebo administered via SC injection (2 injections) q2w starting from Day 1 up to Week 14.
- Placebo - 1 (Open Label): Open-label Treatment Phase: ISB 830 administered at dose of 300 mg (1 × 300 mg) via SC injection q2w starting from Week 16 up to Week 52 (or until participant withdrawal). Participants were followed up for 12 weeks after treatment discontinuation, maximum up to Week 66.
- Placebo - 2 (Blinded): Blinded Treatment Phase: Placebo administered via SC injection (4 injections) q2w starting from Day 1 up to Week 14.
- Placebo - 2 (Open Label): Open-label Treatment Phase: ISB 830 administered at dose of 600 mg (2 × 300 mg) via SC injection q2w starting from Week 16 up to Week 52 (or until participant withdrawal). Participants were followed up for 12 weeks after treatment discontinuation, maximum up to Week 66.
Arm/Group | ISB 830 300 mg q2w | ISB 830 300 mg q4w | ISB 830 75 mg q4w | Placebo - 1 (Blinded) | Placebo - 1 (Open Label) | ISB 830 600 mg q2w | Placebo - 2 (Blinded) | Placebo - 2 (Open Label)
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/78 | 0/77 | 0/80 | 0/60 | 1/75 | 0/74 | 0/67
Serious Adverse Events (participants affected / at risk) | 4/76 | 6/78 | 4/77 | 1/80 | 2/60 | 1/75 | 0/74 | 2/67
Other Adverse Events (participants affected / at risk) | 68/76 | 56/78 | 64/77 | 57/80 | 43/60 | 65/75 | 37/74 | 38/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ISB 830 300 mg q2w (N=76) | ISB 830 300 mg q4w (N=78) | ISB 830 75 mg q4w (N=77) | Placebo - 1 (Blinded) (N=80) | Placebo - 1 (Open Label) (N=60) | ISB 830 600 mg q2w (N=75) | Placebo - 2 (Blinded) (N=74) | Placebo - 2 (Open Label) (N=67)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Eye complication associated with device (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chorioretinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ISB 830 300 mg q2w (N=76) | ISB 830 300 mg q4w (N=78) | ISB 830 75 mg q4w (N=77) | Placebo - 1 (Blinded) (N=80) | Placebo - 1 (Open Label) (N=60) | ISB 830 600 mg q2w (N=75) | Placebo - 2 (Blinded) (N=74) | Placebo - 2 (Open Label) (N=67)
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 6 | 1 | 0 | 3 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0 | 4 | 0 | 0
Fatigue (General disorders) | 2 | 5 | 1 | 0 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 4 | 5 | 1 | 0 | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 16 | 15 | 10 | 7 | 9 | 12 | 7 | 8
Oral herpes (Infections and infestations) | 2 | 3 | 6 | 2 | 4 | 2 | 2 | 3
Sinusitis (Infections and infestations) | 0 | 1 | 2 | 0 | 3 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 12 | 8 | 13 | 4 | 8 | 6 | 5 | 1
Urinary tract infection (Infections and infestations) | 3 | 4 | 4 | 4 | 4 | 3 | 2 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 3 | 0 | 1 | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 4 | 0 | 3 | 2 | 0 | 0
Headache (Nervous system disorders) | 8 | 7 | 4 | 8 | 5 | 6 | 5 | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3 | 1 | 1 | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 2 | 0 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1 | 4 | 3 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 17 | 24 | 21 | 17 | 12 | 26 | 12 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 1 | 0 | 2 | 2 | 1
Hypertension (Vascular disorders) | 5 | 1 | 0 | 0 | 2 | 3 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 2 | 2 | 0 | 2 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Ear swelling (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid margin crusting (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Application site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 1 | 3 | 0 | 0 | 2 | 2 | 1 | 1
Injection site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Injection site induration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Injection site swelling (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Injection site urticaria (General disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 2 | 1 | 2 | 0 | 1 | 0 | 2 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Therapeutic response unexpected (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Allergy to animal (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abscess oral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial blepharitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 0
Chest wall abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Ear lobe infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema herpeticum (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema impetiginous (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Impetigo (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 3 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmic herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0 | 2 | 1 | 2 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 3 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Pyuria (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 2 | 1 | 2 | 1 | 2 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0
Skin bacterial infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Skin candida (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Superinfection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Superinfection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Trichomoniasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 3 | 1 | 1 | 1 | 0 | 1 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0
Acne pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial vulvovaginitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Eczema infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Enterobiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Genital infection female (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Testicular abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transfusion related complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Streptococcus test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary casts present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine ketone body present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Histamine intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Ligamentitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 2 | 0 | 1 | 0 | 2 | 1
Dysaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thoracic spinal cord paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cervix inflammation (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Premature menopause (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine cervix stenosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ovarian disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 1 | 3 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 3 | 0 | 1 | 0 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Solar urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding study results for a period that is mutually agreed upon between the PI and the Sponsor. The sponsor cannot unilaterally extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT03568162/Prot_SAP_000.pdf